CLINICAL TRIAL: NCT06350851
Title: Development of a New Rapid Diagnostic Test to Support Onchocerciasis Elimination
Acronym: Obi1
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Bioaster (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: BA161WP1
Record Dates: First submitted 2024-03-22; First posted 2024-04-05 (Actual); Last update posted 2025-03-07 (Actual); Status verified 2025-03

CONDITIONS: Onchocerciasis; Loiasis; Mansonelliasis; Healthy Volunteers
Keywords: Onchocerca volvulus; Loa loa; Mansonella perstans; Biplex Rapid Diagnostic Test; Neglected Tropical Diseases
MeSH Terms: conditions — Onchocerciasis; Loiasis; Mansonelliasis; Dipetalonema Infections; Neglected Diseases | interventions — Blood Specimen Collection; Defecation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Group1: Control subjects (non-infected with filariasis) (Other): Blood drawing + feces sample collection
  Interventions: Biological: Biological samples collection (blood drawing + feces)
- Group 2: Subjects mono-infected with Onchocerca volvulus (Other): Blood drawing + feces sample collection
  Interventions: Biological: Biological samples collection (blood drawing + feces)
- Group 3: Subjects mono-infected with Loa loa (Other): Blood drawing + feces sample collection
  Interventions: Biological: Biological samples collection (blood drawing + feces)
- Group 4: Subjects mono-infected with Mansonella perstans (alternatively co-infected with Loa loa) (Other): Blood drawing + feces sample collection
  Interventions: Biological: Biological samples collection (blood drawing + feces)

INTERVENTIONS:
Biological: Biological samples collection (blood drawing + feces) — Blood and feces samples will be collected from each volunteer.

SUMMARY:
Onchocerciasis, also known as river blindness, is one of the disease targeted for elimination by the World Health Organization (WHO) in the group of Neglected Tropical Diseases. Existing diagnostic tools for onchocerciasis have limitations that make mapping, epidemiological assessments and verification of elimination of onchocerciasis difficult. It is in this context that WHO, in its 2021-2030 roadmap for onchocerciasis, has identified the development of new diagnostic tests, or the improvement of existing diagnostic tests, as a critical condition for achieving the goal of eliminating onchocerciasis transmission.

To this end, a series of cross-sectional studies will be carried out in Cameroun over a one year period to collect and characterize biological samples for the development and evaluation of a new rapid diagnostic test for onchocerciasis. The study will target individuals aged 18 and over, mono-infected with one of the filarial species Onchocerca volvulus, Loa loa or Mansonella perstans; and non-infected.

At the end of this study, data on the endemicity of onchocerciasis, loiasis and mansonellosis in the selected communities will be updated. More importantly, a new rapid diagnostic test will be developed, which can then be used to monitor the activities of onchocerciasis control programs.

DETAILED DESCRIPTION:
Onchocerciasis, also known as river blindness, stands as the second leading cause of infectious blindness worldwide. According to estimates by the World Health Organization (WHO), approximately 25 million people are infected globally, with another 90 million at risk. Over 99% of these cases occur in Africa, and vision loss affects around 1.15 million individuals. The primary strategy for combating onchocerciasis currently is Community Directed Treatment with Ivermectin (CDTI), requiring a minimum of 80% therapeutic coverage for 10 -15 years.

Areas of West and Central Africa endemic for loiasis and mansonellasis, where ivermectin may trigger severe side effects, pose a significant challenge in the battle against onchocerciasis. Existing diagnostic tools for onchocerciasis have limitations that make mapping, epidemiological assessments and verification of elimination of onchocerciasis difficult. This situation underscores the importance of improving the specificity of onchocerciasis diagnosis to reduce cross-reactivity and false results due to other parasitic helminths in co-endemic regions. It is in this context that WHO, in its 2021-2030 roadmap for onchocerciasis, has identified the development of new diagnostic tests, or the improvement of existing diagnostic tests, as a critical condition for achieving the goal of eliminating onchocerciasis transmission.

To this end, a series of cross-sectional studies will be carried out to build up a bank of well-characterized biological samples for the development and evaluation of a new rapid diagnostic test for onchocerciasis. These studies will take place in the Centre, Littoral, West and South regions of Cameroon over a one year period. The study will target individuals aged 18 and over, mono-infected with one of the filarial species Onchocerca volvulus, Loa loa or Mansonella perstans; and non-infected. The study will begin with a screening phase during which potential participants will be diagnosed for the different filariasis. Following this screening phase, individuals meeting the inclusion criteria will be selected. Once consent has been obtained, blood samples will be taken for test development and validation of the onchocerciasis RDT. In fact, venous blood sample (in a tube containing EDTA) will be taken for each participant, by venipuncture. After collection, the tube(s) containing the blood will be stored in a cooler containing ice and transported to the laboratory within 6 hours of collection. Once at the laboratory, the plasma will be immediately prepared, then aliquoted and stored at -80ºC until transfer to BIOASTER for development and evaluation of the new diagnostic test for onchocerciasis.

At the end of this study, data on the endemicity of onchocerciasis, loiasis and mansonellosis in the selected communities will be updated. More importantly, a new rapid diagnostic test will be developed, which can then be used to monitor the activities of onchocerciasis control programs.

ELIGIBILITY:
Inclusion Criteria:

* Subjects informed of the objectives of the study and who signed a consent form
* Subjects without filariasis (for control subjects), or
* Subjects mono-infected with Onchocerca volvulus, or
* Subjects mono-infected with Loa loa, or
* Subjects mono-infected with Mansonella perstans or alternatively co-infected with Mansonella perstans and Loa loa

Exclusion Criteria:

* Pregnant or breast-feeding women
* Subjects having taken antihelminthic treatment less than 6 months before the inclusion date

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 400 (Estimated)
Dates: Start 2024-04-15 (Actual); Primary Completion 2025-12 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
Evaluation of the performance of the prototype diagnostic test | Up to 52 weeks
  The prototype will be evaluated with all plasma samples in order to determine the dynamic range of the test and the associated variability, as well as its performance in terms of sensitivity and specificity in relation to non-infected samples, and the absence of cross-reactivity with samples infected by Loa loa and Mansonella perstans.

CONTACTS AND LOCATIONS:
Overall Officials: Philippe LEISSNER, Study Director — Bioaster; Joseph KAMGNO, Principal Investigator — ISM (Higher Institute for Scientific and Medical Research)
Locations (1):
- Higher Institute for Scientific and Medical Research, Yaoundé, Cameroon

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Higher Institute for Scientific and Medical research website — https://www.ismcm.org/
- See also: BIOASTER website — https://www.bioaster.org